CLINICAL TRIAL: NCT06475638
Title: Evaluation of Brachial Artery Pulsatility Index As a Predictor of Successful Supraclavicular Block: a Prospective Observational Study
Brief Title: Brachial Artery Pulsatility Index in Supraclavicular Block
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Doctor, Cairo University
Other Study IDs: pulsatility index in SCB
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Brachial Plexus Anesthesia; Diagnostic Accuracy
Keywords: pulsatility index; successful block; resistive index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: brachial artery doppler — brachial artery doppler evaluation before and after supraclavicular block

SUMMARY:
Investigators aimed to evaluated accuracy of brachial artery doppler derived indices such as change in pulsatility index, resistive index, and waveform morphology in predicting successful supraclavicular block

DETAILED DESCRIPTION:
supraclavicular brachial plexus block gives adequate anesthesia and analgesia for arm and hand surgeries. successful block was classically evaluated via assessment of both sensory and motor functions, However this carry disadvantages of subjective assessment including patient cooperation. objective monitors of successful block depend on sympasthetic mediated changes including perfusion index, thermography, and LASER doppler.

However most of these tools depend on complicated technology and special devices.

therefore it was assumed that the use of brachial artery derived indices such as pulsatility index, resistive index, and waveform morphology would provide simple, easy and economic assessment tool for successful supraclavicular brachial plexus block

ELIGIBILITY:
Inclusion Criteria:

- ASA 1 undergoing forearm or hand surgery

Exclusion Criteria:

* patient refusal allergy to local anesthetics fracture humerus Diabetes Melitus peripheral vascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patient, ASA 1 and will receive supraclavicular brachial plexus block for forearm or hand surgery
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-01-11 (Actual); Study Completion 2025-01-11 (Actual)

PRIMARY OUTCOMES:
the change in pulsatility index as a predictor to successful supraclavicular block | baseline and at 5 minutes interval after block for 30 minutes
  the difference between the index before and after the block divided by the index value before the block

SECONDARY OUTCOMES:
change in resistive index as a predictor for successful block | baseline then at 5 minutes interval for 30 minutes
change in waveform morphology as a predictor to successful block | baseline and within 10 minutes of block

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gamo K, Kuriyama K, Higuchi H, Uesugi A, Nakase T, Hamada M, Kawai H. Ultrasound-guided supraclavicular brachial plexus block in upper limb surgery: outcomes and patient satisfaction. Bone Joint J. 2014 Jun;96-B(6):795-9. doi: 10.1302/0301-620X.96B6.31893. PMID 24891581
- [Background] Abdelnasser A, Abdelhamid B, Elsonbaty A, Hasanin A, Rady A. Predicting successful supraclavicular brachial plexus block using pulse oximeter perfusion index. Br J Anaesth. 2017 Aug 1;119(2):276-280. doi: 10.1093/bja/aex166. PMID 28854539
- [Background] Hollenbeck M, Hilbert N, Meusel F, Grabensee B. Increasing sensitivity and specificity of Doppler sonographic detection of renal transplant rejection with serial investigation technique. Clin Investig. 1994 Aug;72(8):609-15. doi: 10.1007/BF00227454. PMID 7819718
- [Background] Uysal AI, Altiparmak B, Korkmaz Toker M, Dinc Elibol F, Karalezli MN, Demirbilek S. Early and late blood flow changes in the brachial artery following brachial plexus block. Minerva Anestesiol. 2020 Sep;86(9):948-956. doi: 10.23736/S0375-9393.20.14309-8. Epub 2020 Jul 1. PMID 32613812
- [Background] Li J, Karmakar MK, Li X, Kwok WH, Ngan Kee WD. Regional hemodynamic changes after an axillary brachial plexus block: a pulsed-wave Doppler ultrasound study. Reg Anesth Pain Med. 2012 Jan-Feb;37(1):111-8. doi: 10.1097/AAP.0b013e318234007e. PMID 22030722
- [Background] Nelson TR, Pretorius DH. The Doppler signal: where does it come from and what does it mean? AJR Am J Roentgenol. 1988 Sep;151(3):439-47. doi: 10.2214/ajr.151.3.439. PMID 2970215